CLINICAL TRIAL: NCT04978701
Title: Dynamic Changes of the Human Microbiome Predict the Risk of Poor Prognosis in Patients With Acute Ischemic Stroke: a Multi-center Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Zhujiang Hospital (Other); Guangdong Yanling Hospital (Unknown); Shenzhen University General Hospital (Other); The First Hospital Of Qiqihar (Unknown); Huzhou Central Hospital (Other); Zhejiang Greentown Cardiovascular Hospital (Other); People's Hospital of Leshan, Sichuan Province (Unknown)
Responsible Party: Principal Investigator, yinjia, Chief Physician, Nanfang Hospital, Southern Medical University
Other Study IDs: NFEC-2021-220
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke, microbiome, prognosis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood plasm；Faeces；Oral swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recent studies have found a close relationship between acute ischemic stroke(AIS) and gut microbiota, but whether the dynamic changes in human microbiome after stroke can predict poor prognosis of stroke remains unclear. Therefore, we planned to explore the predictive value of human microbiome and its metabolites in stroke prognosis through a multicenter cohort study

DETAILED DESCRIPTION:
This study was designed as a prospective, observational, multicenter cohort study. 2000 patients with AIS will be enrolled continuously through multiple centers. Oral swabs, feces (the day after admission, 1 month, 3 months after the onset of disease) and blood samples (the day after admission, 3 months after the onset of disease) will be collected. After the onset of the disease (1 month, 3 months, 6 months and 12 months), outpatient/telephone follow-up will be conducted to evaluate the neurological function scores of the patients, and the recurrence of stroke and other cardio-cerebrovascular events will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Meet the AIS diagnostic criteria;
* Age 18-80;
* Within 7 days of the onset;
* Signing the informed consent, providing relevant medical history and biological specimens.

Exclusion Criteria:

* mRS > score 2 before onset;
* Serious systemic diseases including malignant tumors;
* Hematological diseases and autoimmune diseases;
* ALT or AST > 2 times the upper limit of normal value or severe liver disease;
* Serum creatinine > 1.5 times the upper normal limit or severe nephropathy;
* History of alcoholism, drug abuse, and chemical poisoning (e.g. pesticide poisoning);
* History of intestinal tumor, irritable bowel syndrome or inflammatory bowel disease or confirmed in hospital;
* Antibiotic use within 1 month before admission;
* Fece cannot be obtained within 4 days after admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who met the eligibility criteria for acute ischemic stroke
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale | 3 months after the onset
  An evaluation of neurological deficits
National Institute of Health stroke scale | 3 months after the onset
  An evaluation of neurological deficits
Major ischemic events | within 3 months
  Major ischemic event is defined as ischemic stroke, myocardial infarction, or death from an ischemic vascular event.

SECONDARY OUTCOMES:
modified Rankin Scale | 6 months after the onset
  An evaluation of neurological deficits
National Institute of Health stroke scale | 6 months after the onset
  An evaluation of neurological deficits
Major ischemic events | within 6 months
  Major ischemic event is defined as ischemic stroke, myocardial infarction, or death from an ischemic vascular event.
modified Rankin Scale | 12 months after the onset
  An evaluation of neurological deficits
National Institute of Health stroke scale | 12 months after the onset
  An evaluation of neurological deficits
Major ischemic events | within 12 months
  Major ischemic event is defined as ischemic stroke, myocardial infarction, or death from an ischemic vascular event.

CONTACTS AND LOCATIONS:
Overall Officials: Yin Jia, Master, Principal Investigator — Department of Neurology, NanFang Hospital, Southern Medical University
Locations (1):
- Department of Neurology, NanFang Hospital, Southern Medical University, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No